CLINICAL TRIAL: NCT06199453
Title: The Evaluation of the Effectiveness, Safety and Tolerability of Treatment, Using a Specialized Prostate-specific Membrane Antigen (PSMA) Labeled with Lutetium177, in Patients with Recurrent And/or Metastatic Adenoid Cystic Carcinoma Originating from the Salivary Glands - an Open, Non-commercial Clinical Trial
Brief Title: The Evaluation of the Effectiveness, Safety and Tolerability of Treatment, Using a PSMA-Lu177, in Patients with ACC- an Open, Non-commercial Clinical Trial
Acronym: LuRM_ACC/2023
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuRM_ACC/2023; EU CT 2023-504699-73-00 (Other: EMA)
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Lutetium; Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Treatment will consist of administration of 6 cycles of lutetium (177Lu) vipivotide-tetraxetan with an activity of 200 mCi (7.4 GBq) at intervals of 6 weeks.
  Interventions: Drug: Lutetium (177Lu) vipivotide tetraxetan

INTERVENTIONS:
Drug: Lutetium (177Lu) vipivotide tetraxetan — 6 cycles of lutetium (177Lu) vipivotide-tetraxetan with an activity of 200 mCi (7.4 GBq) at intervals of 6 weeks
  Other Names: Pluvicto 1 000 MBq/mL

SUMMARY:
Non-commercial phase 2 clinical trial to evaluate the effectiveness, safety and tolerability of treatment using prostate-specific membrane antigen (PSMA) labeled with 177Lutetium in patients with recurrence and/or metastases in adenoid cystic carcinoma originating from the salivary glands of the head and neck region.

Patients with PSMA receptor expression confirmed by PET/CT after administration of 68Ga-PSMA I&T will be eligible for treatment.

DETAILED DESCRIPTION:
It is planned to enroll 32 patients diagnosed with non-resectable recurrence and/or dissemination in the course of ACC, whose general condition and life expectancy justify qualification for diagnosis using PSMA 68Ga and treatment with lutetium (177Lu) vipivotide-tetraxetan

The Study assumes the administration of 6 cycles of treatment (lutetium [177Lu] vipivotide-tetraxetan) at 6-week intervals.

If toxicity occurs, the activity of the next dose of the preparation will be modified or its next administration will be delayed by a maximum of 4 weeks.

After completing 6 cycles of therapy, the participant enters the observation phase, which will last until recurrence of the disease is diagnosed or for 2 years after the end of therapy.

ELIGIBILITY:
Inclusion criteria:

* Signing the informed consent form to participate in the study
* Patients with inoperable, locoregionally advanced or metastatic, histopathologically confirmed adenoid cystic carcinoma of salivary gland
* Age over 18 years
* WHO performance status 0 to 2
* PSMA expression confirmed by PET/CT using 68Ga-PSMA;
* Presence of measurable disease according to RECIST 1.1 criteria
* Adequate function of: bone marrow, liver, kidneys:

bone marrow: neutrophils >1500x10^9/L; thrombocytes >150,000x10^9/L, hemoglobin >9 g/dl liver: bilirubin <2xULN; aminotransferases <3xULN (in patients with liver metastases <5xULN) kidney: eGFR >50 ml/min albumin >2.5 mg/ml

* For women of reproductive age: confirmed negative pregnancy test
* The need to use of a highly effective method of contraception

Exclusion criteria:

* Pregnancy or breastfeeding
* Lack of effective contraception during childbearing age
* Patients with metastases to the brain, meninges or heart
* Severe or significant additional diseases in the opinion of the investigator
* Urinary tract obstruction and/or hydronephrosis.
* Concomitant treatment of another cancer
* Myelosuppressive or nuclear treatment later than 4 weeks after qualification
* Previous treatment with 177Lutetium-labeled PSMA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effectiveness of the study treatment | 2 years after the end of treatment
  Objective response rate (ORR) - RECIST 1.1 score in CT examination 2 years after completion of treatment

SECONDARY OUTCOMES:
Assessment of the effectiveness of the study treatment | Time from the date of initiation of the treatment to the disease progression or death
  Progression free survival
Assessment of the effectiveness of the study treatment | Time from the date of initiation of the treatment to death
  Overall survival
Assessment of the effectiveness of the study treatment | Time from the date of initiation of the treatment to the disease progression or death
  Duration of response
Assessment of quality of life | Time from the the date of initiation of treatment to the disease progression or death
  Assessment of quality of life (according to the EORTC QLQ-C30 and EORTC QLQ-H&N43 questionnaire)
Assessment of safety and tolerance | Time from the date of initiation of the treatment to disease progression or death
  Assessment of safety and tolerance of treatment according to Common Terminology Criteria for Adverse Events v. 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: No